CLINICAL TRIAL: NCT04377399
Title: High-dose Vitamin D Supplementation Reduces Inflammation and Improves Microcirculation in Patients With Diabetic Peripheral Neuropathy
Brief Title: High vs Low Dose Vitamin D in Patients With Diabetic Peripheral Neuropathy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federal State Budgetary Institution, V. A. Almazov Federal North-West Medical Research Centre, of the Ministry of Health (Other)
Collaborators: Tameside Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AAAA-A18-118042390157-9
Record Dates: First submitted 2020-04-29; First posted 2020-05-06 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Diabetes Type 2; Diabetic Neuropathies; Vitamin D Deficiency
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Neuropathies; Vitamin D Deficiency | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high dose (Active Comparator): vitamin D (40,000 IU weekly) for 24 weeks
  Interventions: Drug: Vitamin D
- Low dose (Active Comparator): vitamin D (5,000 IU weekly) for 24 weeks
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — Patients will be randomised to receive either high dose vitamin D (40,000 IU weekly) or low dose vitamin D (5,000 IU weekly) for 24 weeks

SUMMARY:
Aim. To assess the effect of different doses of vitamin D supplementation on peripheral neuropathy in patients with type 2 diabetes mellitus (T2DM).

68 patients with T2DM and peripheral neuropathy will be randomized into two treatment groups: cholecalciferol 5,000 IU once/week and cholecalciferol 40,000 IU once/week orally for 24 weeks. Severity of neuropathy (neuropathy symptom score (NSS), neuropathy disability score (NDS), visual analog scale (VAS)), body mass index (BMI), glycated hemoglobin (HbA1c), 25-hydroxycalciferol (25(OH)D), parathyroid hormone (PTH), serum interleukins (IL) 1β, 6 and 10, C-reactive protein, tumor necrosis factor α and microcirculation (MC) parameters assessed before and after treatment. The initial and final indicators of the skin blood flow (M, σ, Kv) and MC parameters after postural and occlusal tests by laser Doppler flowmetry (LDF). Sixteen subjects without diabetes will represent the control group.

DETAILED DESCRIPTION:
It is well known that vitamin D deficiency along with type 2 diabetes mellitus (T2DM) is a modern pandemic. Development of microvascular complications in T2DM worsens both the prognosis and the patients' quality of life. There is increasing evidence of a possible contribution of vitamin D deficiency to the pathogenesis of diabetes and its complications. Large-scale studies have shown 40% increased risk of developing diabetes in individuals with a reduced 25(OH)D level. A recent interventional prospective study demonstrated no decrease in the risk of T2DM development in patients with prediabetes after two-year treatment with 4,000 IU of vitamin D per day. But, some experts suggested that 4,000 IU is not sufficient supplementation dose for patients with already existing impaired glucose metabolism and on the other hand most study participants had normal basal 25(OH)D level. Along with immune-mediated mechanisms, microcirculation deterioration in patients with diabetes has been found to play an important role in the pathogenesis of microvascular complications including peripheral neuropathy (DPN).

It is believed that vitamin D deficiency also plays a role in the progression of DPN. Thus, the correction of vitamin D deficiency in patients with T2DM is becoming increasingly attractive for the prevention and treatment of microvascular complications. However, the question of the required vitamin D dose and the treatment duration remain highly debatable. The aim of this study was to assess the effect of therapy with different doses of cholecalciferol for 24 weeks on clinical manifestations of peripheral neuropathy, inflammatory markers, and parameters of microcirculation in patients with T2DM.

Patients and Methods: Baseline characteristics will be recorded for all patients including Height, weight, BMI, diabetes status and biochemical parameters. All will be repeated at 24 weeks. Blood will be collected after an overnight fast and stored at -20 degrees until analysis.

Patients will be recruited from the Almazov Research centre, St Petersburg, Russia Federation.

68 patients with T2DM and peripheral neuropathy will be randomized into two treatment groups: cholecalciferol 5,000 IU once/week and cholecalciferol 40,000 IU once/week orally for 24 weeks. Severity of neuropathy (neuropathy symptom score (NSS), neuropathy disability score (NDS), visual analog scale (VAS)), body mass index (BMI), glycated hemoglobin (HbA1c), 25-hydroxycalciferol (25(OH)D), parathyroid hormone (PTH), serum interleukins (IL) 1β, 6 and 10, C-reactive protein, tumor necrosis factor α and microcirculation (MC) parameters assessed before and after treatment. The initial and final indicators of the skin blood flow (M, σ, Kv) and MC parameters after postural and occlusal tests by laser Doppler flowmetry (LDF). Sixteen subjects without diabetes will represent the control group.

ELIGIBILITY:
Inclusion Criteria:

* males and females with T2DM aged 18 to 65 years
* diabetes duration ≥5 years,
* HbA1c <9%,
* stable hypoglycemic,
* hypotensive and hypolipidemic therapy
* neurological deficit 4 points and more according to the neuropathy disability score (NDS).

Exclusion Criteria:

* patients with type 1 diabetes
* hypothyroidism
* glomerular filtration rate (GFR) <45 ml/min/1.73 m2
* current and former smokers
* obliterating atherosclerosis
* diabetic foot or Charcot osteoarthropathy
* inflammatory joint diseases
* oncological diseases
* ongoing infectious diseases or in the preceding four weeks
* alcohol and drug addiction
* history of В12 deficiency
* anemia or current therapy with vitamin B12
* regular use of glucocorticoids
* vitamin D supplements
* anticoagulants
* antidepressants
* tricyclic antidepressants
* anticonvulsants
* opiates
* non-steroidal anti-inflammatory drugs
* vasoprotective and microcirculation correctors
* alpha lipoic acid
* group B vitamins.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2020-01-25 (Actual)

PRIMARY OUTCOMES:
Microcirculation | Baseline and 24 weeks
  Assessment of microcirculatory changes using laser doppler

SECONDARY OUTCOMES:
Interleukins | Baseline and 24 weeks
  Serum interleukins (IL) will be determined by enzyme-linked immunosorbent assay (Bio-Rad 680 Microplate Reader, USA) using the appropriate sets of reagents for enzyme immunoassay to determine the concentration of IL-1β (reference values 0-5.0 pg/ml), IL-6 (reference values 0-7.0 pg/ml), IL-10 (reference values 0-9.1 pg/ml), (Vector-Best, Novosibirsk, Russia) compared from baseline
Tumor necrosis factor-α (TNFα) | Baseline and 24 weeks
  Tumor necrosis factor-α (TNFα) will be determined by enzyme-linked immunosorbent assay (Bio-Rad 680 Microplate Reader, USA) using the appropriate sets of reagents for enzyme immunoassay to determine the concentration of TNFα (reference values 0-8.21 pg/ml) (Vector-Best, Novosibirsk, Russia)
Neuropathy disability score | Baseline and 24 weeks
  Using standard scoring systems and questionnaires. Scoring is: Neuropathy disability score (0-10),
Pain score | Baseline and 24 weeks
  Patients will be asked to score pain on a visual analog scale 0-10 with 10 being the worst pain ever
Neuropathic symptom score | Baseline and 24 weeks
  This will be scored using standard questionnaire 0-9

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana Karonova, PhD, Principal Investigator — Almazov National Medical Research Centre
Locations (1):
- Almazov National Medical Research Centre, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No